CLINICAL TRIAL: NCT03128502
Title: Assessment of Pentraxin-3 Levels in Gingival Crevicular Fluid and Saliva in Periodontal Health and Disease
Brief Title: Estimation of Pentrexin-3 Levels in GCF and Saliva of Patients With Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Professor of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University., Cairo University
Other Study IDs: PTX-3_AgP_CP
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis
Keywords: saliva; GCF; pentraxin-3
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — salivary and GCF samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy control: Ten healthy control subjects presented with clinically healthy periodontium. Control subjects had to meet the following criteria for inclusion: probing depth less than 3mm, no clinical attachment loss, no bleeding on probing, with Gingival and Plaque index 0-1.
- plaque induced gingivitis: Ten patients who had plaque induced gingivitis characterized by the presence of any of the following clinical signs: redness and edema of the gingival tissue, bleeding upon provocation, changes in contour and consistency, presence of calculus and/or plaque, with no clinical attachment loss nor radiographic evidence of bone loss.
- chronic periodontitis: Ten chronic moderate to severe periodontitis patients selected according to the criteria currently adopted by Armitage 1999. Moderate destruction is generally characterized by periodontal probing depths up to 6 mm with clinical attachment loss of up to 4 mm. Advanced destruction is generally characterized by periodontal probing depths greater than 6 mm with attachment loss greater than 4 mm. Radiographic evidence of bone loss is apparent, Increased tooth mobility may be present.
- aggressive periodontitis: Ten patients suffering generalized aggressive periodontitis, patients were less than 35 years of age and had generalized interproximal attachment loss affecting at least 3 permanent teeth other than the first molars and incisors with at least one site each with PD and CAL >5 mm, Attachment loss occurs in pronounced episodic periods of destruction, and there is familial aggregation (subjects were asked if they had at least one other member of the family presenting or with a history of periodontal diseases).

SUMMARY:
Subjects were selected from the outpatient clinic, Department of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University. Ten healthy control subjects presented with clinically healthy periodontium. Ten patients who had plaque induced gingivitis. Ten patients who had generalized chronic periodontitis. Ten patients who had generalised aggressive periodontitis. Pentraxin-3 levels were evaluated in GCF and saliva of all subjects included in this study with ELISA technique.

DETAILED DESCRIPTION:
The study population consisted of 4 groups of forty patients selected as follows:

Group 1 - Healthy Controls:

Ten healthy control subjects presented with clinically healthy periodontium. Control subjects had to meet the following criteria for inclusion: probing depth less than 3mm, no clinical attachment loss, no bleeding on probing, with Gingival and Plaque index 0-1.

Group 2 - Plaque induced gingivitis patients:

Ten patients who had plaque induced gingivitis characterized by the presence of any of the following clinical signs: redness and edema of the gingival tissue, bleeding upon provocation, changes in contour and consistency, presence of calculus and/or plaque, with no clinical attachment loss nor radiographic evidence of bone loss.

Group 3 - Chronic periodontitis group:

Ten chronic moderate to severe periodontitis patients selected according to the criteria currently adopted by Armitage 1999. Moderate destruction is generally characterized by periodontal probing depths up to 6 mm with clinical attachment loss of up to 4 mm. Advanced destruction is generally characterized by periodontal probing depths greater than 6 mm with attachment loss greater than 4 mm. Radiographic evidence of bone loss is apparent, Increased tooth mobility may be present.

Group 4 - Aggressive periodontitis group:

Ten patients suffering generalized aggressive periodontitis, patients were less than 35 years of age and had generalized interproximal attachment loss affecting at least 3 permanent teeth other than the first molars and incisors with at least one site each with PD and CAL >5 mm, Attachment loss occurs in pronounced episodic periods of destruction, and there is familial aggregation (subjects were asked if they had at least one other member of the family presenting or with a history of periodontal diseases).

GCF and saliva samples were collected for all patients. Pentraxin-3 levels were evaluated in GCF and saliva of all subjects included in this study with ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

* patients with plaque induced gingivitis
* patients with chronic periodontitis
* patients with aggressive periodontitis

Exclusion Criteria:

* Patients with any systemic disease according to Cornell medical index (1968).
* Patients taking any medications or antibiotics in the last 3 months.
* Current or former smoker patients.
* Pregnant females.

Ages: 25 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients from the outpatient clinic, Department of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University suffering from diffrent periodontal diseases.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
GCF and salivary pentraxin-3 levels | baseline
  levels of pentraxin-3 in GCF and saliva

SECONDARY OUTCOMES:
plaque index | baseline
  Oral hygiene status of the patients were recorded using the plaque index of Silness & Lӧe (1964)
gingival index | baseline
  Performed using the gingival index of Lӧe (1967)
probing pocket depth | baseline
  The depths of the periodontal pockets were measured as the distance from the gingival margin to the base of the pocket using periodontal probe with William's graduation.
clinical attachment level | baseline
  Clinical attachment levels were measured as the distance from the CEJ to the base of the pocket using William's graduated periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Engy Ahmed, M.D., Study Director — Associate Professor of Oral Medicine & Periodontology, faculty of Oral and Dental Medicine, Cairo University; Yasmine Mansour, B.D.Sc, Principal Investigator — master candidate at faculty of dentistry cairo university; Olfat Shaker, Study Chair — Professor of Medical Biochemistry, Faculty of Medicine, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fujita Y, Ito H, Sekino S, Numabe Y. Correlations between pentraxin 3 or cytokine levels in gingival crevicular fluid and clinical parameters of chronic periodontitis. Odontology. 2012 Jul;100(2):215-21. doi: 10.1007/s10266-011-0042-1. Epub 2011 Sep 20. PMID 21932007
- [Result] Lakshmanan R, Jayakumar ND, Sankari M, Padmalatha O, Varghese S. Estimation of pentraxin-3 levels in the gingival tissues of chronic and aggressive periodontitis participants: an in vivo study. J Periodontol. 2014 Feb;85(2):290-7. doi: 10.1902/jop.2013.120718. Epub 2013 May 23. PMID 23701480
- [Result] Gumus P, Nizam N, Nalbantsoy A, Ozcaka O, Buduneli N. Saliva and serum levels of pentraxin-3 and interleukin-1beta in generalized aggressive or chronic periodontitis. J Periodontol. 2014 Mar;85(3):e40-6. doi: 10.1902/jop.2013.130281. Epub 2013 Aug 16. PMID 23952075